CLINICAL TRIAL: NCT04081766
Title: Randomized Controlled Trial of Pharmacist-Led Patient Counselling in Controlling Hypoglycemic Attacks in Older Adults With Type 2 Diabetes Mellitus
Brief Title: Pharmacist-Led Study in Controlling Hypoglycemia in Older Adults With Type 2 Diabetes Mellitus
Acronym: ROSE-ADAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lincoln (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-May-0170
Record Dates: First submitted 2019-09-04; First posted 2019-09-09 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2020-11

CONDITIONS: Diabetes Mellitus Type 2 With Hypoglycemia
Keywords: Diabetes Mellitus, Type 2; Diabetes Mellitus; Hypoglycemia; Counseling; Older Adults
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SUGAR Handshake (Active Comparator): Participants assigned to the intervention group will receive an individualised, pharmacist-led patient counselling session (SUGAR Handshake package) at the inclusion visit.
  Participants will also receive a pictogram with the main instructions for easy recall of the counselling contents.
  They will also receive a glucometer and test strips with a demonstration on proper use, to measure their fasting blood glucose levels on a daily basis for 12 weeks.
  At week 6, participants will receive a phone call to reinforce the intervention and to remind them of the study protocol. For the qualitative evaluation of the intervention, a number of participants are interviewed and asked questions through the sixth week-phone call.
  Additionally, participants in this group will be provided with the usual care that is normally provided in the outpatient clinics at King Abdullah University Hospital.
  Interventions: Behavioral: SUGAR Handshake
- Control (No Intervention): Participants within this group will receive the usual care provided by the health care professionals in the outpatient clinics at King Abdullah University Hospital.
  They will also be provided with instructions on hypoglycemia diagnosis, and treatment and a demonstration on glucometer use at the inclusion visit. They will be asked to measure their fasting blood glucose level daily for 12 weeks.
  Participants will receive a phone call at week 6 of the inclusion visit to remind them of measuring blood glucose levels and documenting hypoglycemic episodes on the diaries., plus a counselling session about hypoglycaemia recognition and treatment at the inclusion visit.
  For the qualitative evaluation of the study, a number of participants will be interviewed and asked questions through the sixth week-phone call.

INTERVENTIONS:
Behavioral: SUGAR Handshake — An interactive patient counselling session delivered by a pharmacist which mainly focuses on medication-related instructions towards preventing hypoglycaemia in addition to recommendations about hypoglycemia early recognition, causes, and treatment. The SUGAR Handshake is individualised according to shared decision making and each participant's characteristics.
  Components of the SUGAR Handshake intervention will be covered under five main domains:
  1. Signs and symptoms of hypoglycemia.
  2. Understanding the underlying causes of hypoglycaemia such as misuse of anti-diabetic medications.
  3. Good glycaemic control and self-monitoring, which mainly includes instructions on handling the anti-diabetic medications.
  4. Acknowledgement by the patient
  5. Recap and summary
  The pictogram contains the main recommendations for easy recall by the participant. Moreover, the intervention will be reinforced by a phone call at week 6 of the inclusion visit.
  Arms: SUGAR Handshake

SUMMARY:
This study involves two parts: a randomised controlled trial, and a nested qualitative study.

The main aim of the trial is to evaluate the effectiveness of a pharmacist-led, medications-focused patient counselling on reducing the frequency of hypoglycaemia in older adults diagnosed with type 2 Diabetes Mellitus within 12 weeks in Jordan.

The study hypothesis is that individualised patient counselling which is provided by pharmacists and involves recommendations about anti-diabetic medications will reduce the risk of hypoglycaemia by preventing further episodes in the elderly Jordanians with type 2 Diabetes Mellitus.

The qualitative study aims at evaluating the experience of participants in both groups with the study (process evaluation). This involves exploring which components are effective and which are not with the reasons, the contextual factors affecting the delivery and implementation of the study and the intervention, and how the study and the intervention can be scaled up in the future.

DETAILED DESCRIPTION:
Hypoglycaemia is the most serious adverse effect of diabetes treatment. Older adults are at the highest risk to develop hypoglycaemia. Several studies have established the important positive role of educational interventions on achieving glycaemic control and other clinical outcomes, however, there is still a lack in clinical trials that evaluate the impact of such type of interventions on hypoglycaemia risk, especially in older adults. Despite the increasing prevalence of chronic diseases such as diabetes in Jordan, pharmacists still provide traditional services rather than patient-centred services.

The purpose of this research is to investigate the effect of pharmacist-led, individualised, and medications-focused patient counselling on reducing episodes of hypoglycaemia compared to the usual care in older Jordanians with type 2 Diabetes Mellitus within 12 weeks.

This research is a prospective, open-label, randomised controlled trial that is conducted in the outpatient endocrinology and cardiology clinics at King Abdullah University Hospital in Jordan, with 204 elderly patients who had been diagnosed with type 2 diabetes. Participants will be randomised in a 1:1 ratio into either the intervention (SUGAR Handshake) or the usual care groups. Each participant in the SUGAR Handshake group will receive a face-to-face individualised educational session with a pharmacist at the inclusion visit, a pictogram containing the main educational information, and a reinforcement of the educational session through a phone call at week 6 of the inclusion visit. They will also receive the usual care provided by the health care professionals at the outpatient clinics. On the other hand, patients in the usual care group will only receive the routine care provided at the outpatient clinics. The duration of the trial for each participant is 12 weeks.

The qualitative study is performed through phone interviews with 8-12 participants of each group at week 6 of the inclusion visit. Participants are to be approached according to convenience sampling and the data will be analysed using content analysis.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of type 2 Diabetes Mellitus
* Have been taking a sulfonylurea, insulin, or any three or more anti-diabetic medications

Exclusion Criteria:

* Unable to understand instructions or to give consent.
* Impaired mental capacity
* On palliative care for cancer, with advanced-stage or end-stage diseases, who have psychosis or severe depression, who are terminally-ill, or with life expectancy < 6 months
* Have been diagnosed with haemolytic anaemia or hemoglobinopathies as being self-reported or according to the patient's electronic record.
* Unwilling to take home glucose measurements or to use the glucometer (for example because of severe hearing or visual impairment and without a caregiver to measure the blood glucose level by the glucometer)
* Unwilling to return for follow up.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 212 (Actual)
Dates: Start 2020-02-09 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Frequency of total episodes of hypoglycaemia | 12 weeks
  The frequency of hypoglycemia will be calculated as the number of total hypoglycemic episodes/person/ 12 weeks. Total hypoglycemia is defined as the summation of severe, symptomatic, and asymptomatic episodes of hypoglycaemia.

SECONDARY OUTCOMES:
Frequency of severe hypoglycaemia | 12 weeks
  The frequency of severe hypoglycemia will be calculated as the number of severe hypoglycemic episodes/person/ 12 weeks. Severe hypoglycemia is defined as any event requiring the assistance of another person to administer carbohydrate and glucagon or take any other corrective actions, accompanied by neurological recovery after the corrective actions.
  Participants will be provided with diaries to document severe episodes of hypoglycemia
Frequency of asymptomatic hypoglycemia | 12 weeks
  The frequency of asymptomatic hypoglycemia will be calculated as the number of asymptomatic hypoglycaemia episodes/person/ 12 weeks. asymptomatic hypoglycaemia is defined as an event not accompanied by typical symptoms of hypoglycemia but with a measured plasma glucose concentration ≤70 mg/dL (≤3.9 mmol/L).
  Participants will be provided with diaries to document fasting blood glucose levels by which asymptomatic episodes will be diagnosed.
Frequency of symptomatic hypoglycemia | 12 weeks
  The frequency of symptomatic hypoglycemia will be calculated as the number of symptomatic hypoglycemic episodes/person/ 12 weeks. Symptomatic hypoglycemia is defined as an event during which the patient experiences typical symptoms of hypoglycaemia (sweating, dizziness, light-headedness, tremor, hunger, headache) whether they are accompanied by a measured plasma glucose concentration ≤70 mg/dL (≤3.9 mmol/L) or not.
  Participants will be provided with diaries to document symptomatic episodes of hypoglycemia.
Proportion of patients experiencing hypoglycaemia | 12 weeks
  proportion of patients who experience at least one hypoglycaemic attack of each type
Time to the first hypoglycaemic attack | 12 weeks
  the number of the day when a participant will experience the first hypoglycaemic attack of any type after randomisation.

CONTACTS AND LOCATIONS:
Overall Officials: Keivan Ahmadi, PhD, Study Director — Associate Professor in Pharmacology & Therapeutics, Lincoln Medical School
Locations (1):
- King Abdullah University Hospital, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Almomani HY, Ayre HM, Powell RA, Armani K. The SUGAR handshake intervention to prevent hypoglycaemia in elderly people with type 2 diabetes: process evaluation within a pragmatic randomised controlled trial. BMC Geriatr. 2025 Oct 1;25(1):753. doi: 10.1186/s12877-025-06361-2. PMID 41034834
- [Derived] Almomani HY, Pascual CR, Al-Azzam SI, Ahmadi K. Randomised controlled trial of pharmacist-led patient counselling in controlling hypoglycaemic attacks in older adults with type 2 diabetes mellitus (ROSE-ADAM): A study protocol of the SUGAR intervention. Res Social Adm Pharm. 2021 May;17(5):885-893. doi: 10.1016/j.sapharm.2020.07.012. Epub 2020 Jul 29. PMID 32763086